CLINICAL TRIAL: NCT04431271
Title: Retrospective Comparative Study on Costs of Conventional Versus Robotic Assisted Laparoscopic Groin Hernia Repair
Brief Title: Economic Assessment of STarting Endoscopic Robotic Groin Hernia Repair
Acronym: EASTER
Status: Completed | Type: Observational
Sponsor: Algemeen Ziekenhuis Maria Middelares (Other)
Responsible Party: Principal Investigator, Filip Muysoms, Principal Investigator, Algemeen Ziekenhuis Maria Middelares
Other Study IDs: EASTER study
Record Dates: First submitted 2020-06-05; First posted 2020-06-16 (Actual); Last update posted 2020-08-27 (Actual); Status verified 2020-08

CONDITIONS: Inguinal Hernia
MeSH Terms: conditions — Hernia, Inguinal

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Robot-assisted laparoscopy: Patients who underwent robot-assisted groin hernia repair
  Interventions: Procedure: Robot-assisted hernia repair
- Conventional laparoscopy: Patients who underwent conventional laparoscopic groin hernia repair

INTERVENTIONS:
Procedure: Robot-assisted hernia repair — Inguinal hernia repair was performed using the DaVinci Xi robotic system
  Groups: Robot-assisted laparoscopy

SUMMARY:
The material cost for robotic groin hernia repair is higher than for conventional laparoscopic surgery. In this study, this amount will be quantified and possible differences in early postoperative course, hospital stay and readmission rate that could influence the cost/benefit ratio for robotic groin hernia surgery will be analyzed.

DETAILED DESCRIPTION:
Robot-assisted groin hernia repair has been introduced in AZ Maria Middelares hospital since September 2016. In these procedures, the daVinci robot is being used to perform minimal invasive repair of these hernias. At the moment, this technique is frequently being used for groin hernia repair. Literature shows a clear benefit of robot-assisted versus open repair. Hospital stay decreases and complications are less frequently observed in patients who underwent minimal invasive repair (Henriksen NA et al., 2018).

On the other hand, the benefits of robot-assisted repair are less obvious compared to conventional laparoscopy. Many robot-trained surgeons are in favor of robot-assisted repair, but current literature is still inconclusive about the economic feasibility of robot-assisted groin hernia repair as standard of care.

This retrospective observational study is primarily designed to analyze the additional cost of robot-assisted groin hernia repair compared to conventional laparoscopic repair. A cost-benefit analysis will be carried out for groin hernia repairs performed by the same surgeon (Dr. Filip Muysoms) in the period 2016-2019.

As primary endpoint, direct costs related to the introduction of robot-assisted groin hernia repair will be analyzed. These are: material costs, costs related to hospital stay, honoraria and costs related to intrahospital complications. A comparison will be made between conventional laparoscopic and robot-assisted groin hernia repair.

As secondary endpoint, indirect costs will be compared between both groups. These include costs related to late complications and readmissions related to the index operation.

ELIGIBILITY:
Inclusion Criteria:

* adult patients
* underwent uni-or bilateral groin hernia repair in the period 2015- 2019
* surgery through minimal invasive repair

Exclusion Criteria:

* open surgery or conversion from minimal-invasive to open surgery
* combined procedures
* age below 18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients who underwent uni-or bilateral groin hernia repair in the period 2015- 2019. Only patients who underwent minimal-invasive surgery (conventional or robot-assisted laparoscopy) will be included.
Sampling Method: Non-Probability Sample
Enrollment: 677 (Actual)
Dates: Start 2020-06-01 (Actual); Primary Completion 2020-07-31 (Actual); Study Completion 2020-07-31 (Actual)

PRIMARY OUTCOMES:
Direct costs | Immediately post hospital discharge
  Material costs, hospitalization costs, specialist fees and costs related to early complications

SECONDARY OUTCOMES:
Indirect costs | 0- 42 days postoperatively
  Late complication costs, readmission costs

CONTACTS AND LOCATIONS:
Overall Officials: Filip Muysoms, MD, PhD, Principal Investigator — Algemeen Ziekenhuis Maria Middelares
Locations (1):
- AZ Maria Middelares, Ghent, Oost-Vlaanderen, Belgium